CLINICAL TRIAL: NCT00910507
Title: The Impact of Physical Therapist-Directed Exercise Counseling Combined With Fitness Center-Based Exercise Training on Stage of Exercise Behavior in People With Type 2 Diabetes: A Randomized Clinical Trial
Brief Title: The Impact of Exercise Counseling on Exercise Behavior in People With Type 2 Diabetes: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Arkansas (Other)
Responsible Party: James David Taylor, PT, PhD (Principal Investigator), University of Central Arkansas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCA IRB 07-070
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2009-06-01 (Estimated); Status verified 2009-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Exercise; Counseling; Behavior
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise counseling (Experimental): Each participant in the experimental group receives exercise counseling from the same physical therapist as described in previous research. In short, during each exercise counseling session, the physical therapist addresses the benefits of exercise for people with type 2 diabetes, advises each participant to adhere to the prescribed exercise program, and assists each participant by reviewing the prescribed exercise program. Exercise counseling is tailored to the stage of exercise behavior as described in previous literature. The experimental group is also provided access to a fitness center.
  Interventions: Behavioral: Exercise counseling
- Supervised exercise training (Active Comparator): Participants who are randomly allocated to the comparison group receive a 2-month supervised exercise program. Each participant in the comparison group receives the same prescribed exercise program as the experimental group and is supervised during each exercise training session by a trained co-investigator in a controlled exercise laboratory setting.
  Interventions: Behavioral: Supervised exercise training

INTERVENTIONS:
Behavioral: Exercise counseling — Each participant in the experimental group receives 2 months of exercise counseling from the same physical therapist as described in previous research. In short, during each exercise counseling session, the physical therapist addresses the benefits of exercise for people with type 2 diabetes, advises each participant to adhere to the prescribed exercise program, and assists each participant by reviewing the prescribed exercise program. Exercise counseling is tailored to the stage of exercise behavior as described in previous literature. The experimental group is also provided access to a fitness center.
  Arms: Exercise counseling
Behavioral: Supervised exercise training — Participants who are randomly allocated to the comparison group receive a 2-month supervised exercise program. Each participant in the comparison group receives the same prescribed exercise program as the experimental group and is supervised during each exercise training session by a trained co-investigator in a controlled exercise laboratory setting.
  Arms: Supervised exercise training

SUMMARY:
The purpose of this randomized clinical trial is to investigate the impact of physical therapist-directed exercise counseling combined with fitness center-based exercise training on stage of exercise behavior in people with type 2 diabetes.

DETAILED DESCRIPTION:
Type 2 diabetes is a chronic, metabolic disease characterized by hyperglycemia resulting from insulin resistance. Research studies indicate that complications such as cardiovascular disease, peripheral vascular disease, retinopathy, and loss of physical function are associated with type 2 diabetes. Clinical management of people with type 2 diabetes consists of medical nutrition therapy, pharmacological therapy, and exercise. Exercise has been shown to improve risk factors associated with complications of type 2 diabetes such as elevated plasma glucose, elevated blood pressure, loss of muscular strength, and loss of exercise capacity. In fact, the American Diabetes Association and American College of Sports Medicine have published position statements recommending the use of exercise, specifically resistance and aerobic training, as an intervention for people with type 2 diabetes. However, 31 percent of people with type 2 diabetes have reported no regular physical activity and an additional 38 percent have reported less than recommended levels of physical activity. Therefore, interventions to promote regular exercise behavior in people with type 2 diabetes are clinically important by potentially preventing type 2 diabetes-related complications.

Previous studies have investigated the impact of exercise counseling on exercise behavior in people with type 2 diabetes. However, these studies have limitations such as lack of agreement with exercise training guidelines for people with type 2 diabetes and research design flaws. This current study investigates the effect of a novel, physical therapist-directed exercise counseling combined with fitness center-based exercise training intervention on stage of exercise behavior in people with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Consider medically stable to participate by a physician

Exclusion Criteria:

* Contraindication for exercise testing
* Uncontrolled hypertension
* Proliferative retinopathy
* Severe peripheral neuropathy
* Nephropathy
* Autonomic neuropathy
* Unable to participate due to a physical impairment
* Fasting plasma glucose greater than 250 mg/dL
* Involved in resistance or aerobic training on 2 or more days per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Stage of Exercise Behavior | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: James D Taylor, PT, PhD, Principal Investigator — University of Central Arkansas
Locations (1):
- University of Central Arkansas, Conway, Arkansas, United States